# **Study Protocol with Statistical Analysis Plan**

# **Study Title**

The Effectiveness of Wearable Devices on Health Promotion in Individuals with Diabetes Mellitus

# **Principal Investigator**

Eliza Wu, PT, PhD Doctor of Physical Therapy Program Pacific University

Email: eliza.wu@pacificu.edu | Phone: 503-352-7259



# Proposal to Conduct Research

| Institutional Review Board<br>FWA: 00007392 IRB: 0004173 |
|------------------------------------------------------------|
| 2032697-1 |
| IRB Number |
| 09/14/2023 |
| Approved |
| 12/01/2023 |
| Post-Approval Request(s) |
| 09/14/2024 |
| Approval Expires |

# 1. Study Objectives

This randomized controlled pilot study aims to evaluate the effectiveness of wrist-worn activity trackers (Fitbit Inspire 2) on improving physical activity levels, cardiovascular risk factors, and quality of life in adults diagnosed with type 2 diabetes over a 4-week period.

# 2. Study Design

- Type: Interventional (Clinical Trial), two-arm parallel design

- Randomization: Yes (1:1 allocation)

Blinding: NoneDuration: 4 weeks

- Sample Size: 20 participants (10 per group)

# 3. Eligibility Criteria

Inclusion Criteria:

- Age ≥ 18 years
- Diagnosed with type 2 diabetes (HbA1c ≥ 6.5% or fasting glucose ≥ 126 mg/dL)
- Willing and able to link a fitness tracker app to a smartphone

#### **Exclusion Criteria:**

- Use of assistive devices for walking
- Current smokers
- Pregnant or breastfeeding
- Already achieving ≥150 min/week of moderate-to-vigorous activity
- Comorbidities preventing participation in physical activity
- Current insulin therapy

# 4. Intervention and Control Groups

Intervention Group: Participants receive a Fitbit Inspire 2.

Control Group: Participants do not receive a wearable device.

### 5. Outcome Measures

**Primary Outcomes:** 

- Physical activity: Measured using Global Physical Activity Questionnaire (GPAQ) and pedometer/mobile app data
- Cardiovascular risk: Measured using arterial stiffness (SphygmoCor), blood pressure, heart rate, fasting glucose, BMI, waist-to-hip ratio

### Secondary Outcomes:

- Health-related quality of life: Measured using the RAND SF-36 Health Survey

# 6. Statistical Analysis

Descriptive statistics will summarize baseline characteristics. Non-parametric tests will be used:

- Friedman's test and Wilcoxon signed-rank tests (within-group change)
- Mann–Whitney U test (between-group comparison)
- Spearman's rho for correlations

Effect sizes (r) will be calculated. All analyses will be conducted using IBM SPSS v29. Significance set at p < 0.05.

# 7. Data Management and Confidentiality

Data will be stored in a secure BOX folder regulated by the PI. No identifiable data will be stored on local or personal devices. Data will be retained for five years post-study.

### 8. Risks and Benefits

Risks: Minimal; primarily related to fasting and physical exertion.

Benefits: Participants may gain insight into their physical activity levels and cardiovascular health.

Compensation: None, though participants in the intervention group may retain their Fitbit upon study completion.

#### 9. Ethical Considerations

IRB Approval: Pacific University IRB #2032697-1

Informed consent is obtained electronically via Qualtrics in English or Spanish. No deception is used. Adverse events will be monitored and reported per IRB policy.

### 10. Timeline

- Recruitment: Upon IRB approval
- Data Collection: Week 0 (T0) and Week 4 (T1)
- Analysis & Dissemination: Expected completion within 3 months post-data collection